CLINICAL TRIAL: NCT01296399
Title: The Rate of In-stent Restenosis Within Bare Metal Stents as Compared to Drug Eluting Stents in Patients With Patent Previously Deployed Bare Metal Stent
Brief Title: In-stent Restenosis in Patients With Patent Previous Bare Metal Stent
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Dr. Doron Sudarsky, Rambam Medical Center
Other Study IDs: 02511CTIL
Record Dates: First submitted 2011-02-13; First posted 2011-02-15 (Estimated); Last update posted 2011-02-15 (Estimated); Status verified 2011-02

CONDITIONS: In-stent Coronary Artery Restenosis
Keywords: in stent restenosis; bare metal stent; drug eluting stent; de novo lesion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Bare metal stent: patients, with a patent previously deployed intra coronary bare metal stent, receiving intra coronary bare metal stent, for de-novo stenosis
- Drug eluting stent: patients, with a patent previously deployed intra coronary bare metal stent, receiving intra coronary drug eluting stent, for de-novo stenosis

SUMMARY:
Intra-coronary stents deployment reduces the rate of angiographic restenosis as compared to Balloon angioplasty. in-stent restenosis, usually defined as ≥50 percent diameter stenosis within previously deployed stent, is most often becoming clinically evident within the first 6 to 12 months after the stent was deployed. Several risk factors are predictors for the development of in-stent restenosis. These can be generally calcified as either clinical, angiographic or procedural related factors. However it is difficult to estimate to what extent In stent re-stenosis is influenced by these various components.

Drug eluting stent, as compared to bare metal stents, markedly reduced the incidence of angiographic in-stent restenosis. However this benefit must be weighed against a suggested increased risk of late and very late stent thrombosis, a catastrophic event often leading to myocardial infarction and death. Often in patients with existing risk factors for in-stent restenosis, drug eluting stents will be deployed even in cases where patency of a previously deployed bare metal stent have been demonstrated.

Therefore the researchers sought to investigate whether in patients with previously deployed bare metal stent and no evidence of in-stent re-stenosis there will be a significant difference in the rates of in-stent between drug eluting stents and bare metal stents deployed within de-novo stenotic lesions.

DETAILED DESCRIPTION:
Intra-coronary stents deployment reduces the rate of angiographic restenosis and clinically-driven repeat target lesion revascularization (TLR) compared to percutaneous transluminal coronary angioplasty (PTCA) alone. Angiographic binary in-stent restenosis (ISR) is usually defined as ≥50 percent diameter stenosis within previously deployed intra-coronary stent. in-stent restenosis is most often becoming clinically evident within the first 6 to 12 months after the stent was deployed. Although there is an increase in neointimal tissue with subsequent reduction in the minimal luminal diameter (MLD) during the first six months after stent deployment, there may be no further reduction in luminal diameter, or even regression, at one year and a further increase in diameter at later time points. Hence, after one year recurrent ischemia is more likely to be due to new or progressive disease at another site rather than due to ISR.

Several risk factors are predictors for the development of ISR. These can be generally calcified as clinical related factors, angiographic related factors and procedural related factors:

clinical related factors- higher rates of ISR are seen in female patients, hypertensive or diabetic patients , patients suffering from multivessel disease or renal dysfunction and stenting performed in the setting of acute coronary syndrome (ACS).

angiographic related factors -higher rates of ISR are seen in some lesion types, such as smaller reference artery diameter, Smaller pretreatment MLD, longer lesion length, complex lesions, ostial lesions, ISR in a companion lesion or stenting of multiple lesions and bifurcation lesions and treatment of in-stent restenosis.

procedural related factors- lower rates of ISR are seen after high-pressure post-dilation while higher rates of ISR are seen with stent under-expansion, placement of multiple stents, longer stent length (>35 mm) and stented segment, Excessive stent length in relation to the lesion length, Overlapping stents, smaller post-treatment MLD (MLD after stenting <3 mm), post-procedural percent diameter residual stenosis, the use of coil stent and a shorter time interval, between prior angioplasty and current stent implantation. The configuration of the stent may also affect ISR rates. Stents with thinner strut thickness are less likely to demonstrate ISR. Contact allergy to metal compounds, particularly nickel, released from stainless steel stents have also been suggested to contribute to the development of ISR.

Drug eluting stents (DES) demonstrate the ability to suppress in-stent neointimal hyperplasia, a sustained effect that lasts even after two years from the time the DES was deployed. Multiple randomized trials, large registries and meta-analyses have demonstrated that drug DES, as compared to bare metal stents (BMS), markedly reduced the incidence of angiographic in-stent restenosis (ISR), rates of late lumen loss as well as the rates of target lesion revascularization (TLR).Likely scenarios, both "on-label" and "off label" use, for the preference of DES over BMS, owing to improved efficacy, include stenosis of the Left main coronary artery, left main equivalent disease, and stenosis of the ostial or proximal left anterior descending artery, large amount of viable myocardium at risk, need for multi-vessel revascularization, long lesions, stenosis of small diameter vessels, complex or bifurcation lesions, restenotic lesions, saphenous vein graft stenosis and chronic total occlusion (CTO). In most North America centers, DES have been utilized in preference to BMS whenever feasible.However the benefits of DES on ISR must be weighed against the concerns in regard to the suggested increased risk of late and very late stent thrombosis, especially if dual antiplatelet therapy with aspirin and a thienopyridine is prematurely discontinued, a catastrophic event often leading to myocardial infarction and death.Furthermore, the longer time period recommended with dual antiplatelet treatment, after deployment of DES as compared to BMS, poses an increased risk of major bleeding.

There is an increase in the use of DES. In patients suffering from ISR in other arteries or other segments of the artery, DES will often be deployed in de-novo stenotic lesions. However, it is difficult to estimate to what extent ISR is influenced by the various predictors for ISR. in patients with either clinical angiographic or procedural related risk factors, DES will often be deployed even in cases where patency of a previously deployed BMS have been demonstrated. Therefore the researchers sought to investigate whether in patients with previously deployed BMS and no evidence of ISR, so-called "non-restenosers", there will be a significant difference in the rates of ISR between DES and BMS deployed within de-novo stenotic lesions.

ELIGIBILITY:
Inclusion Criteria:

* The patient underwent coronary angiography and subsequent angioplasty with deployment of a bare metal stent within de novo stenotic lesion.
* The patient underwent a second coronary procedure, more then six month from the first procedure, in which patency of the previously deployed bare metal stent was demonstrated, provided that no intervention was performed within this stent in the six month interim. In lieu, either bare metal stent or drug eluting stent were deployed within another stenotic lesion (another de novo lesion).
* The patient underwent a third coronary angiography procedure within the 12 month interim from the second coronary procedure, in which in-stent restenosis was demonstrated within the stent deployed in the second procedure
* If no in-stent restenosis was demonstrated within the stent, deployed in the second procedure within the 12 month interim from the second procedure, the patient underwent coronary angiography at least 12 month from the second procedure in which patency of the bare metal stent or drug eluting stent was determined

Exclusion Criteria:

* Patients in whom a stent, in either the first or second procedure was deployed within previously stent treated stenotic lesion.
* Patients in whom a stent, in either the first or second procedure, was deployed within a graft.
* Patient suffering from in-stent restenosis within the bare metal stent, during the six month interim between the first procedure and second procedure or at the time of the second coronary angiography
* Patients who underwent a coronary intervention within the bare metal stent in interim between the first and second procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients who underwent percutaneous coronary intervention in Rambam Medical Center between 2000 -2010.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2000-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The rate of angiographic in-stent restenosis of a stent deployed within de-novo lesions | one year after the stent was deployed

SECONDARY OUTCOMES:
all cause mortality all cause mortality | one year after the stent was deployed

CONTACTS AND LOCATIONS:
Overall Officials: Doron Sudarsky, MD, Principal Investigator — Rambam Health Care Campus; Arthur Kerner, MD, Study Chair — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel

REFERENCES:
- [Background] Serruys PW, de Jaegere P, Kiemeneij F, Macaya C, Rutsch W, Heyndrickx G, Emanuelsson H, Marco J, Legrand V, Materne P, et al. A comparison of balloon-expandable-stent implantation with balloon angioplasty in patients with coronary artery disease. Benestent Study Group. N Engl J Med. 1994 Aug 25;331(8):489-95. doi: 10.1056/NEJM199408253310801. PMID 8041413
- [Background] Fischman DL, Leon MB, Baim DS, Schatz RA, Savage MP, Penn I, Detre K, Veltri L, Ricci D, Nobuyoshi M, et al. A randomized comparison of coronary-stent placement and balloon angioplasty in the treatment of coronary artery disease. Stent Restenosis Study Investigators. N Engl J Med. 1994 Aug 25;331(8):496-501. doi: 10.1056/NEJM199408253310802. PMID 8041414
- [Background] Cutlip DE, Chauhan MS, Baim DS, Ho KK, Popma JJ, Carrozza JP, Cohen DJ, Kuntz RE. Clinical restenosis after coronary stenting: perspectives from multicenter clinical trials. J Am Coll Cardiol. 2002 Dec 18;40(12):2082-9. doi: 10.1016/s0735-1097(02)02597-4. PMID 12505217
- [Background] Goldberg SL, Loussararian A, De Gregorio J, Di Mario C, Albiero R, Colombo A. Predictors of diffuse and aggressive intra-stent restenosis. J Am Coll Cardiol. 2001 Mar 15;37(4):1019-25. doi: 10.1016/s0735-1097(01)01107-x. PMID 11263602
- [Background] Cutlip DE, Chhabra AG, Baim DS, Chauhan MS, Marulkar S, Massaro J, Bakhai A, Cohen DJ, Kuntz RE, Ho KK. Beyond restenosis: five-year clinical outcomes from second-generation coronary stent trials. Circulation. 2004 Sep 7;110(10):1226-30. doi: 10.1161/01.CIR.0000140721.27004.4B. Epub 2004 Aug 30. PMID 15337693
- [Background] Kornowski R, Hong MK, Tio FO, Bramwell O, Wu H, Leon MB. In-stent restenosis: contributions of inflammatory responses and arterial injury to neointimal hyperplasia. J Am Coll Cardiol. 1998 Jan;31(1):224-30. doi: 10.1016/s0735-1097(97)00450-6. PMID 9426044
- [Background] Komatsu R, Ueda M, Naruko T, Kojima A, Becker AE. Neointimal tissue response at sites of coronary stenting in humans: macroscopic, histological, and immunohistochemical analyses. Circulation. 1998 Jul 21;98(3):224-33. doi: 10.1161/01.cir.98.3.224. PMID 9697822
- [Background] Kimura T, Yokoi H, Nakagawa Y, Tamura T, Kaburagi S, Sawada Y, Sato Y, Yokoi H, Hamasaki N, Nosaka H, et al. Three-year follow-up after implantation of metallic coronary-artery stents. N Engl J Med. 1996 Feb 29;334(9):561-6. doi: 10.1056/NEJM199602293340903. PMID 8569823
- [Background] Kuroda N, Kobayashi Y, Nameki M, Kuriyama N, Kinoshita T, Okuno T, Yamamoto Y, Komiyama N, Masuda Y. Intimal hyperplasia regression from 6 to 12 months after stenting. Am J Cardiol. 2002 Apr 1;89(7):869-72. doi: 10.1016/s0002-9149(02)02205-1. No abstract available. PMID 11909579
- [Background] Hoffmann R, Mintz GS. Coronary in-stent restenosis - predictors, treatment and prevention. Eur Heart J. 2000 Nov;21(21):1739-49. doi: 10.1053/euhj.2000.2153. No abstract available. PMID 11052838
- [Background] Kastrati A, Schomig A, Elezi S, Schuhlen H, Dirschinger J, Hadamitzky M, Wehinger A, Hausleiter J, Walter H, Neumann FJ. Predictive factors of restenosis after coronary stent placement. J Am Coll Cardiol. 1997 Nov 15;30(6):1428-36. doi: 10.1016/s0735-1097(97)00334-3. PMID 9362398
- [Background] Lemos PA, Hoye A, Goedhart D, Arampatzis CA, Saia F, van der Giessen WJ, McFadden E, Sianos G, Smits PC, Hofma SH, de Feyter PJ, van Domburg RT, Serruys PW. Clinical, angiographic, and procedural predictors of angiographic restenosis after sirolimus-eluting stent implantation in complex patients: an evaluation from the Rapamycin-Eluting Stent Evaluated At Rotterdam Cardiology Hospital (RESEARCH) study. Circulation. 2004 Mar 23;109(11):1366-70. doi: 10.1161/01.CIR.0000121358.26097.06. Epub 2004 Mar 1. PMID 14993127
- [Background] Singh M, Gersh BJ, McClelland RL, Ho KK, Willerson JT, Penny WF, Holmes DR Jr. Clinical and angiographic predictors of restenosis after percutaneous coronary intervention: insights from the Prevention of Restenosis With Tranilast and Its Outcomes (PRESTO) trial. Circulation. 2004 Jun 8;109(22):2727-31. doi: 10.1161/01.CIR.0000131898.18849.65. Epub 2004 Jun 1. PMID 15173022
- [Background] Kastrati A, Schomig A, Elezi S, Dirschinger J, Mehilli J, Schuhlen H, Blasini R, Neumann FJ. Prognostic value of the modified american college of Cardiology/American heart association stenosis morphology classification for long-term angiographic and clinical outcome after coronary stent placement. Circulation. 1999 Sep 21;100(12):1285-90. doi: 10.1161/01.cir.100.12.1285. PMID 10491372
- [Background] Kastrati A, Schomig A, Elezi S, Schuhlen H, Wilhelm M, Dirschinger J. Interlesion dependence of the risk for restenosis in patients with coronary stent placement in in multiple lesions. Circulation. 1998 Jun 23;97(24):2396-401. doi: 10.1161/01.cir.97.24.2396. PMID 9641690
- [Background] Kobayashi Y, De Gregorio J, Kobayashi N, Akiyama T, Reimers B, Finci L, Di Mario C, Colombo A. Stented segment length as an independent predictor of restenosis. J Am Coll Cardiol. 1999 Sep;34(3):651-9. doi: 10.1016/s0735-1097(99)00303-4. PMID 10483943
- [Background] Savage MP, Fischman DL, Rake R, Gebhardt S, Goldberg S. Interprocedural interval as a predictor of stent restenosis after previous coronary angioplasty. The Palmaz-Schatz Stent Investigators. Am J Cardiol. 1996 Sep 15;78(6):683-4. doi: 10.1016/s0002-9149(96)00397-9. PMID 8831408
- [Background] Castagna MT, Mintz GS, Leiboff BO, Ahmed JM, Mehran R, Satler LF, Kent KM, Pichard AD, Weissman NJ. The contribution of "mechanical" problems to in-stent restenosis: An intravascular ultrasonographic analysis of 1090 consecutive in-stent restenosis lesions. Am Heart J. 2001 Dec;142(6):970-4. doi: 10.1067/mhj.2001.119613. PMID 11717599
- [Background] Mauri L, O'Malley AJ, Popma JJ, Moses JW, Leon MB, Holmes DR Jr, Teirstein PS, Cutlip DE, Donahoe D, Kuntz RE. Comparison of thrombosis and restenosis risk from stent length of sirolimus-eluting stents versus bare metal stents. Am J Cardiol. 2005 May 15;95(10):1140-5. doi: 10.1016/j.amjcard.2005.01.039. PMID 15877983
- [Background] Costa MA, Simon DI. Molecular basis of restenosis and drug-eluting stents. Circulation. 2005 May 3;111(17):2257-73. doi: 10.1161/01.CIR.0000163587.36485.A7. No abstract available. PMID 15867193
- [Background] Aoki J, Colombo A, Dudek D, Banning AP, Drzewiecki J, Zmudka K, Schiele F, Russell ME, Koglin J, Serruys PW; TAXUS II Study Group. Peristent remodeling and neointimal suppression 2 years after polymer-based, paclitaxel-eluting stent implantation: insights from serial intravascular ultrasound analysis in the TAXUS II study. Circulation. 2005 Dec 20;112(25):3876-83. doi: 10.1161/CIRCULATIONAHA.105.558601. Epub 2005 Dec 12. PMID 16344384
- [Background] Roiron C, Sanchez P, Bouzamondo A, Lechat P, Montalescot G. Drug eluting stents: an updated meta-analysis of randomised controlled trials. Heart. 2006 May;92(5):641-9. doi: 10.1136/hrt.2005.061622. Epub 2005 Oct 10. PMID 16216853
- [Background] Moses JW, Leon MB, Popma JJ, Fitzgerald PJ, Holmes DR, O'Shaughnessy C, Caputo RP, Kereiakes DJ, Williams DO, Teirstein PS, Jaeger JL, Kuntz RE; SIRIUS Investigators. Sirolimus-eluting stents versus standard stents in patients with stenosis in a native coronary artery. N Engl J Med. 2003 Oct 2;349(14):1315-23. doi: 10.1056/NEJMoa035071. PMID 14523139
- [Background] Stettler C, Wandel S, Allemann S, Kastrati A, Morice MC, Schomig A, Pfisterer ME, Stone GW, Leon MB, de Lezo JS, Goy JJ, Park SJ, Sabate M, Suttorp MJ, Kelbaek H, Spaulding C, Menichelli M, Vermeersch P, Dirksen MT, Cervinka P, Petronio AS, Nordmann AJ, Diem P, Meier B, Zwahlen M, Reichenbach S, Trelle S, Windecker S, Juni P. Outcomes associated with drug-eluting and bare-metal stents: a collaborative network meta-analysis. Lancet. 2007 Sep 15;370(9591):937-48. doi: 10.1016/S0140-6736(07)61444-5. PMID 17869634
- [Background] Iakovou I, Ge L, Colombo A. Contemporary stent treatment of coronary bifurcations. J Am Coll Cardiol. 2005 Oct 18;46(8):1446-55. doi: 10.1016/j.jacc.2005.05.080. Epub 2005 Sep 28. PMID 16226167
- [Background] Schofer J, Schluter M, Gershlick AH, Wijns W, Garcia E, Schampaert E, Breithardt G; E-SIRIUS Investigators. Sirolimus-eluting stents for treatment of patients with long atherosclerotic lesions in small coronary arteries: double-blind, randomised controlled trial (E-SIRIUS). Lancet. 2003 Oct 4;362(9390):1093-9. doi: 10.1016/S0140-6736(03)14462-5. PMID 14550694
- [Background] Ardissino D, Cavallini C, Bramucci E, Indolfi C, Marzocchi A, Manari A, Angeloni G, Carosio G, Bonizzoni E, Colusso S, Repetto M, Merlini PA; SES-SMART Investigators. Sirolimus-eluting vs uncoated stents for prevention of restenosis in small coronary arteries: a randomized trial. JAMA. 2004 Dec 8;292(22):2727-34. doi: 10.1001/jama.292.22.2727. PMID 15585732
- [Background] Stone GW, Ellis SG, Cannon L, Mann JT, Greenberg JD, Spriggs D, O'Shaughnessy CD, DeMaio S, Hall P, Popma JJ, Koglin J, Russell ME; TAXUS V Investigators. Comparison of a polymer-based paclitaxel-eluting stent with a bare metal stent in patients with complex coronary artery disease: a randomized controlled trial. JAMA. 2005 Sep 14;294(10):1215-23. doi: 10.1001/jama.294.10.1215. PMID 16160130
- [Background] Williams DO, Abbott JD, Kip KE; DEScover Investigators. Outcomes of 6906 patients undergoing percutaneous coronary intervention in the era of drug-eluting stents: report of the DEScover Registry. Circulation. 2006 Nov 14;114(20):2154-62. doi: 10.1161/CIRCULATIONAHA.106.667915. Epub 2006 Oct 23. PMID 17060386
- [Background] Ong AT, Hoye A, Aoki J, van Mieghem CA, Rodriguez Granillo GA, Sonnenschein K, Regar E, McFadden EP, Sianos G, van der Giessen WJ, de Jaegere PP, de Feyter P, van Domburg RT, Serruys PW. Thirty-day incidence and six-month clinical outcome of thrombotic stent occlusion after bare-metal, sirolimus, or paclitaxel stent implantation. J Am Coll Cardiol. 2005 Mar 15;45(6):947-53. doi: 10.1016/j.jacc.2004.09.079. PMID 15766834
- [Background] Ong AT, McFadden EP, Regar E, de Jaegere PP, van Domburg RT, Serruys PW. Late angiographic stent thrombosis (LAST) events with drug-eluting stents. J Am Coll Cardiol. 2005 Jun 21;45(12):2088-92. doi: 10.1016/j.jacc.2005.02.086. PMID 15963413
- [Background] Iakovou I, Schmidt T, Bonizzoni E, Ge L, Sangiorgi GM, Stankovic G, Airoldi F, Chieffo A, Montorfano M, Carlino M, Michev I, Corvaja N, Briguori C, Gerckens U, Grube E, Colombo A. Incidence, predictors, and outcome of thrombosis after successful implantation of drug-eluting stents. JAMA. 2005 May 4;293(17):2126-30. doi: 10.1001/jama.293.17.2126. PMID 15870416